CLINICAL TRIAL: NCT06859944
Title: Prospective Randomized Non-Inferiority Study Comparing Natural Cycle Frozen Embryo Transfer (NC-FET) to a New Type of Endometrial Preparation for FET: Natural Proliferative Phase (NPP-FET)
Acronym: NPP
Status: Recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Anne Delbaere, Professor, Erasme University Hospital
Other Study IDs: SRB2024108
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Comparison of Pregnancy Rate (HCG+ Level) Obtained After a Replacement Embryonic in Spontaneous Cycle and Following Protocol "NPP". Comparison
MeSH Terms: interventions — Embryo Transfer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- single transfer of frozen blastocyst in natural cycle
  Interventions: Other: Embryo transfer
- Natural Cycle Programmed by Progesterone
  Interventions: Other: Embryo transfer

INTERVENTIONS:
Other: Embryo transfer — Frozen embryo transfer
  Groups: Natural Cycle Programmed by Progesterone
Other: Embryo transfer — Frozen Embryo transfer
  Groups: single transfer of frozen blastocyst in natural cycle

SUMMARY:
Frozen embryo replacement cycle :Two methods traditionally used: the spontaneous cycle and the artificial cycle.Now, Emergence of new protocols: NPP-FET or "Natural proliferative phase - frozen embryo transfer" Demonstrate non-inferiority between the NPP-FET and the spontaneous cycle, and superiority in terms of planning.

DETAILED DESCRIPTION:
The protocol Natural proliferative phase/Natural Programmed by Progesterone, Patients with regular cycles, candidates for replacement of embryos frozen in a spontaneous cycle. The monitoring of the cycle is carried out by taking blood and follicular ultrasound between the 10th and 13th day of the cycle. Support luteal phase by intravaginal progesterone (utrogestan 200 mg) 1 tablet, 2 times per day, is initiated once the following criteria are met:

* Thickness of the endometrium > 7 mm on ultrasound
* Ovarian follicle > 14 mm
* Estradiol( E2) > 120 pg/mL Embryo transfer is scheduled on the 6th day of progesterone exposure exogenous. A progesterone dosage on the day of transfer will be systematically realized

ELIGIBILITY:
Inclusion Criteria:

* Single transfer Blastocyste

Exclusion Criteria:

* PGT (Preimplantation genetic diagnosis)
* Testicular Sperm
* Donor oocytes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Patients with regular cycles, candidates for replacement of embryos frozen in spontaneous cycle
Study Population: Patients with regular cycles, candidates for replacement of embryos frozen in spontaneous cycle
Sampling Method: Probability Sample
Enrollment: 272 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the pregnancy rate (Human chorionic gonadotropin hormone) (HCG+ level) obtained after spontaneous embryo replacement and following the "NPP" protocol. | Thrugh study completion (9 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No